CLINICAL TRIAL: NCT03674528
Title: Technical Validation of Magnetic Resonance Biomarkers of Obesity-Associated Non-Alcoholic Fatty Liver Disease
Brief Title: Technical Validation of MR Biomarkers of Obesity-Associated NAFLD
Acronym: NAFLD
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); GE Healthcare (Industry); Pfizer (Industry); Siemens Medical Solutions (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0244; 2R01DK088925-06A1 (NIH); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 3/8/2022 (Other: UW Madison); 5UL1TR002373-04 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2018-09-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: MRI; MRE; Liver Disease; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group: Subjects with a BMI of 35 or more will be asked to undergo a single MRE imaging session.
  Interventions: Other: Magnetic Resonance Elastography (MRE)
- Patient Group: Adults that are candidates for weight loss surgery will be asked to participate in four study visits that include MRE imaging and 1 - 2 liver biopsy procedures.
  Interventions: Other: Magnetic Resonance Elastography (MRE); Diagnostic Test: Liver biopsy

INTERVENTIONS:
Other: Magnetic Resonance Elastography (MRE) — The MRE scan will several breath holds and will take approximately 30 minutes to complete.
  Other Names: MRI
Diagnostic Test: Liver biopsy — Subjects undergoing WLS will be asked to allow for liver biopsy samples to be collected during their surgical procedure. The collection of these samples will take approximately 5 minutes to complete.
  Other Names: Intraoperative Biopsy
  Groups: Patient Group

SUMMARY:
The overall goal of this collaborative research program is to develop, validate and translate advanced quantitative magnetic resonance (MR) biomarkers of obesity-associated non-alcoholic fatty liver disease (NAFLD). This protocol represents the research plan for two distinct phases. The first phase is an optimization phase. The second phase is designed to complete a rigorous test of conventional and advanced MRE techniques. Complementary anthropometric, laboratory, and MR measures will also be collected to characterize the cohort and identify factors that affect MRE performance

DETAILED DESCRIPTION:
The long-term objective of this research is to improve the health of the millions of Americans with or at risk for NAFLD, the most common chronic liver disease and most rapidly growing indication for liver transplantation in the United States. To achieve this objective, an advanced MR-based imaging method will be used to measure liver "stiffness" which is an early sign of disease. This technique has been previously developed and validated and ready to be used for further research. This current protocol will extend previous work by optimizing and validating advanced 2 dimensional and 3 dimensional-magnetic resonance elastography (MRE) methods as non-invasive biomarkers of hepatic inflammation and fibrosis in obese patients at risk for non-alcoholic steatohepatitis (NASH), the histologically more aggressive subset of NAFLD.

Per Amendment approved 4/8/22: MRE exams will be conducted using a PDFF Pocket Phantom purchased by the UCSD from Calimetrix. This phantom consists of vials with known fat fraction which are captured when taking images of the liver. The known fat fractions provide an independent reference and are used for quality assurance purposes.

ELIGIBILITY:
Inclusion Criteria (Phase 1 and 2 participants)

* Age of at least 18 years
* Severely obese (BMI ≥ 35 kg/m2) patient

Inclusion Criteria (Phase 2 participants only)

* Cleared for weight-loss surgery
* Willing and able to complete all safety and follow-up procedures
* Willing to allow for the banking of biological samples

Exclusion Criteria (Phase 1 and 2 participants)

* Contraindications to MRI
* Girth or weight that exceeds scanner capacity
* Women of childbearing potential that are pregnant or will be attempting to become pregnant during the study duration.

Exclusion Criteria (Phase 2 participants only)

* Known liver malignancies
* Regular & excessive alcohol consumption within 2 years prior to recruitment
* Use of steatogenic or hepatotoxic drugs
* Clinical or laboratory evidence of liver disease other than Nonalcoholic fatty liver disease (NAFLD)/ Nonalcoholic steatohepatitis (NASH) (e.g. HCV Ab, HBV Ab, ceruloplasmin)
* The subject has increased bleeding risk (i.e., decreased platelets, von Willebrand disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase 1 participants will be healthy adults with a BMI of greater/equal to 35 kilograms per meter squared.
  Phase 2 participants must be eligible for weight loss surgery and willing to undergo a liver biopsy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Optimization of MRE for 2 dimensional and 3 dimensional methods | Up to 24 months
  Optimize MRE wave-field generation in this subject population to maximize the area of invertible shear waves in the liver into interpretable shear stiffness maps.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reeder, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - University of Wisconsin, Madison, Madison, Wisconsin